CLINICAL TRIAL: NCT06593626
Title: A Phase I Clinical Study on the Safety and Pharmacokinetics of [18F]Florbetazine Injection in Healthy Subjects and Patients With Amyloid Fibrils
Brief Title: A Phase I Clinical Study on the Safety and Pharmacokinetics of [18F]Florbetazine Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HTA Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YZGK-FBZ-Ι-001
Record Dates: First submitted 2024-05-24; First posted 2024-09-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-09

CONDITIONS: MCI; AD
Keywords: 18F; MCI; AD; phase Ⅰ

STUDY DESIGN:
Intervention Model Description: Single-center, multi-dose, open-dosing study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- [18F]Florbetazine, 10mCi (Experimental): Evaluate the safety and pharmacokinetics of [18F]Florbetazine injection in healthy subjects.
  Interventions: Drug: [18F]Florbetazine
- [18F]Florbetazine, 10mCi, 8mCi, 5mCi (Experimental): AD and MCI
  Interventions: Drug: [18F]Florbetazine

INTERVENTIONS:
Drug: [18F]Florbetazine — Evaluate the safety of [18F]Florbetazine injection in AD and MCI patients, and healthy subjects.

SUMMARY:
This study is a phase-1 study that aims to evaluate the safety and pharmacokinetics of [18F]Florbetazine injection in healthy subjects and patients with MCI and AD.

This study has evaluated and compared the distributed patterns of [18F]Florbetazine injection in healthy subjects and patients with AD and MCI.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects

  1. Male and Female subjects aged 50-85 years (including 50 ang 85 years);
  2. Fertile men or women must use effective birth control during the study period (effective contraception means sterilization, intrauterine hormonal devices, condoms, contraceptives/pills, abstinence or excision vas deferens, etc.) For healthy subjects

  <!-- -->

  1. Sign informed consent;
  2. Good health status or no major diseases are judged by the researcher based on the following assessments: medical history, health results of vital signs, physical examination, clinical electrocardiogram and clinical laboratory examination;
  3. Normal blood routine, blood biochemistry, urine routine and coagulation routine during the screening period, or abnormal without clinical significance;
  4. According to neuropsychological tests and researchers' judgment, no cognitive impairment;
  5. The score of clinical dementia rating (CDR) is 0;
  6. The score of mini-mental state examination (MMSE) is equal or greater than 27; For MCI patients

  <!-- -->

  1. Sign informed consent;
  2. Diagnosed as Alzheimer's disease-related mild cognitive impairment (AD-MCI) according to the diagnostic criteria of NIA-AA;
  3. The Aβ-PET imaging displays positive result;
  4. The score of clinical dementia rating (CDR) is 0.5;
  5. The score of mini-mental state examination (MMSE) is equal or less than 27; For AD patients

  <!-- -->

  1. Sign informed consent;
  2. According to NIA-AA clinical criteria, the patients could be diagnosed as AD dementia;
  3. The Aβ-PET imaging displays positive result;
  4. Mild to moderate dementia, and the score of clinical dementia rating (CDR) is 1 or 2;
  5. The score of mini-mental state examination (MMSE) is 10-17 (illiteracy), or 10-22 (primary school graduate), or 10-24 (middle school graduate), or 10-26 (college and above graduate), the score with upper and lower limits.
  6. Caregivers who live with the patient or regularly look after the patient are willing to provide information about the patient's cognitive status

Exclusion Criteria:

* For all subjects

  1. Pregnant (positive pregnancy test during screening) or breastfeeding women;
  2. A history of alcohol or drug abuse/dependence;
  3. Known allergies to radiation and alcohol, or other severe allergies;
  4. Human immunodeficiency virus (HIV), hepatitis C virus (HCV) or treponema pallidum antibody test positive, hepatitis B virus (HBV) surface antigen positive;
  5. A history of liver disease or other conditions that interfere with drug absorption, distribution, excretion, or metabolism as determined by the investigator;
  6. Blood clotting history or blood clotting disorder;
  7. The subject has cognitive impairment due to causes other than AD, including but not limited to: a. Injuries caused by acute or post-traumatic brain injury, subdural hematoma, or chronic trauma: e.g. boxing sequelae; b. Hypoxic brain injury (regardless of cause) : cognitive or neurological impairment, such as cardiac arrest or cardiac surgery, anesthesia, or severe autotoxic episodes secondary to severe hypovolemia (orthostatic hypotension does not result in exclusion of subjects); c. Confirm vitamin deficiency status based on medical history: such as folic acid, vitamin B12 and other B complex vitamins deficiency; Such as vitamin B1 deficiency in Korsakoff syndrome (note: subjects taking regular B12 and folic acid do not necessarily need to be excluded); d. Brain infections, including abscesses, syphilis, meningitis, encephalitis, or AIDS; e. Primary or metastatic brain tumors; f. Toxic diseases, such as chronic alcoholism, organic poisoning, CO poisoning; g. Significant endocrine or metabolic diseases such as thyroid, parathyroid or pituitary diseases, Cushing's syndrome or severe renal failure; h. Mental retardation;
  8. The subject has clinically significant infarction or possible multiple infarct dementia, including: a. A history of significant cerebrovascular events leading to physical or neurological impairment, which may affect the assessment of the subject's intellectual function; b. Neurological examination showed a variety of focal signs of the nervous system, suggesting multiple ischemic attacks; (1) Multiple (2 or more) infarcts or critical site infarcts: a large (>1.5 cm in diameter) infarct in the area of the cerebral angular gyrus, thalamus, basal forebrain, posterior cerebral artery (PCA), or anterior cerebral artery (ACA); ② Widespread periventricular white matter disease. A distinction needs to be made between leukoosteoporosis (periventricular white matter, low attenuation) and multiple cerebral infarction. Leukoosteoporosis is a common condition in the normal population and in Alzheimer's disease. Leukodegeneration will not result in exclusion of subjects unless it is abnormal and widespread, as in Binswanger disease.
  9. The present presence of clinically significant mental illness based on medical history, especially the present presence of major depression or schizophrenia;
  10. A history of epilepsy or convulsions, but not febrile convulsions in childhood;
  11. Significant occupational exposure to ionizing radiation (e.g., more than 50 MSV/year) within the past 10 years;
  12. Unable to repeat venipuncture;
  13. Have had metal devices implanted that are not compatible with MR, including pacemakers or defibrillators, insulin pumps, cochlear implants, intraocular metal implants, nerve stimulators, CNS aneurysm clips, etc., or have claustrophobia or cannot tolerate imaging procedures for other reasons;
  14. received any drug or treatment before enrollment that the investigator determines may interfere with the trial data or may cause serious side effects and is not fully eluted;
  15. Participating in other drug clinical studies and using other investigational drugs within 30 days prior to screening;
  16. Subjects received radiopharmaceutical imaging or treatment within 7 days prior to screening;
  17. Other conditions that the investigator considers inappropriate to participate in the clinical trial; For healthy subjects

  <!-- -->

  1. Have a history of dementia or other genetic history;
  2. Meet the criteria for MCI or dementia diagnosis, or have been diagnosed before;
  3. Have been on medication for cognitive impairment or dementia;
  4. Any previous major illness or unstable condition (e.g. unstable angina pectoris, dilated or hypertrophic cardiomyopathy, valvular heart disease, congenital heart disease, myocardial infarction or coronary revascularization, heart failure, chronic kidney failure, chronic liver disease, severe lung disease, blood disease, diabetes, chronic infection, epilepsy, mental illness); For AD patients

  <!-- -->

  1. Have received a non-vaccine investigational treatment for Alzheimer's disease or other dementias within the last 3 months (or 5 half-lives of the drug, whichever is older), or have received a passive immunotherapy drug (antibody) used to treat Alzheimer's disease or other dementias within the last 6 months, or have previously received a vaccine used to treat Alzheimer's disease or other dementias;
  2. Have neurodegenerative diseases other than Alzheimer's disease, including but not limited to: Parkinson's disease, Pick's disease, frontotemporal degeneration (FTLD), Huntington's disease, Down's syndrome, Creutzfeldt-Jakya disease, normal pressure hydrocephalus, and progressive suprachinuclear palsy (PSP);
  3. Have been or are currently diagnosed with dementia other than AD, including but not limited to Parkinson's disease dementia, Lewy body dementia, frontotemporal dementia, vascular dementia, mixed dementia, etc.;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events (AE) and their incidence during the trial, | 30 day
  Safety and tolerability: Adverse events (AE) and their incidence during the trial, clinical symptoms and signs (including vital signs), laboratory findings.

SECONDARY OUTCOMES:
Standard uptake value ratio | The whole process from collection to follow-up trial was completed
  Evaluation of the standard uptake value ratio (SUVR) of [18F]Florbetazine injection in the regions of interesting (ROI), and the whole cerebellum is regarded as reference region.
Bio-distribution | The whole process from collection to follow-up trial was completed
  At different time points after drug injection, perform PET/CT whole-body scans to obtain radioactivity counts (%ID) in major irradiated organs at each phase, reflecting the drug's biodistribution in the body.
Multi-dose exploration | The whole process from collection to follow-up trial was completed
  PET/CT scan images, including measuring the standardized uptake value (SUV) within the integrated region of interest (iROI), subjective assessment of image quality, to evaluate the impact of drug dose on image quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Pan M, Yu H, Zhang Q, Chang Y, Zhao H, Wang J, Wang X, Dai J, Yu L, Chen D, Zhang J, Yan XX, Yao S, Cui M. Preclinical and preliminary clinical evaluation of [18F]Florbetazine for non-invasive PET detection of cardiac amyloidosis. Eur J Nucl Med Mol Imaging. 2026 Jan 10. doi: 10.1007/s00259-025-07719-9. Online ahead of print. PMID 41518400